CLINICAL TRIAL: NCT02007603
Title: Multiple-dose Pharmacokinetics of Ampicillin / Sulbactam and Amoxicillin / Clavulanic Acid During Haemodialysis in Longterm Haemodialysis Patients
Brief Title: Concentration of Ampicillin / Sulbactam and Amoxicillin / Clavulanic Acid in the Blood During Renal Replacement Therapy in Longterm Renal Replacement Therapy Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Florian Thalhammer, a.o.Univ.-Prof. Dr., Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AMPISUL/AMOXICLAV-HD_V1.4
Record Dates: First submitted 2013-10-16; First posted 2013-12-11 (Estimated); Last update posted 2017-05-31 (Actual); Status verified 2017-05

CONDITIONS: Infection During Hemodialysis
Keywords: chronic hemodialysis; ampicillin; sulbactam; amoxicillin; clavulanic acid; pharmacokinetics
MeSH Terms: interventions — Clavulanic Acid; sultamicillin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ampicillin / sulbactam (Experimental): Patients are randomized to the ampicillin / sulbactam arm. Pharmacokinetic samples will be taken during multiple hemodialysis sessions.
  Interventions: Drug: Ampicillin / sulbactam; Procedure: Blooddraws for pharmacokinetic profiling
- Amoxicillin / clavulanic acid (Experimental): Patients are randomized to the amoxicillin / clavulanic acid arm. Pharmacokinetic samples will be taken during multiple hemodialysis sessions.
  Interventions: Drug: Administration of Amoxicillin / clavulanic acid; Procedure: Blooddraws for pharmacokinetic profiling

INTERVENTIONS:
Drug: Administration of Amoxicillin / clavulanic acid — Patients receive amoxicillin / clavulanic acid due to clinical necessity
  Arms: Amoxicillin / clavulanic acid
Drug: Ampicillin / sulbactam — Patients receive ampicillin / sulbactam due to clinical necessity
  Arms: Ampicillin / sulbactam
Procedure: Blooddraws for pharmacokinetic profiling — Blood will be sampled at multiple timepoints during multiple hemodialysis sessions

SUMMARY:
The study will be conducted to investigate the pharmacokinetics of ampicillin / sulbactam and amoxicillin/clavulanic acid during intermittent haemodialysis.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Suspected or proven bacterial infection requiring parenteral antibiotic therapy.
* Renal replacement therapy (HD)

Exclusion Criteria:

* Known hypersensitivity to ampicillin / sulbactam, amoxicillin / clavulanic acid or other beta-lactames, or severe hypersensitivity (anaphylactic reaction) to beta-lactam antibacterial agents.
* An expected survival of less than two days.
* Known pregnancy
* Co-administration of one of the following drugs: probenecid which cannot be discontinued for the duration of the study
* Ampicillin / sulbactam respectively amoxicillin / clavulanic acid as monotherapy for resistant species or fungal infections.
* Other reasons opposing the study participation on the discretion of the investigators.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2013-08 (Actual); Primary Completion 2015-02 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Influence of hemodialysis on the area under concentration curve of ampicillin/sulbactam and amoxicillin / clavulanic acid plasma concentration levels. | day 15
  Pharmacokinetic samples are drawn on multiple timepoints from each patient during his participation.

CONTACTS AND LOCATIONS:
Overall Officials: Florian Thalhammer, Prof. MD, Principal Investigator — Medical University of Vienna
Locations (1):
- Medical University of Vienna, Vienna, Austria